CLINICAL TRIAL: NCT03011723
Title: Positive Emotions, Communication and Quality of Life in Dementia: A Tailored Music Therapy Intervention
Brief Title: Tailored Music Therapy for Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: NKS Olaviken Alderspsykiatriske sykehus (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UBergen 2016/1374
Record Dates: First submitted 2016-12-12; First posted 2017-01-05 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer Dementia; Dementia, Vascular; Dementia, Lewy Body; Dementia Parkinson's Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular; Lewy Body Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Music therapy (Experimental): 10 weekly sessions of in-home music therapy for PWDs and a caregiver, including weekly practicing of the interventions with the caregiver between the sessions. The treatment is administered individually.
  Interventions: Behavioral: Resource oriented music therapy

INTERVENTIONS:
Behavioral: Resource oriented music therapy — 10 weeks of tailored individual music therapy for PWD and a caregiver. Pre and post assessment in addition.
  The music therapy consists of one or more of the following activities:
  1. Singing
  2. Listening to live music
  3. Listening to recorded music
  4. Dancing
  5. Conversations about memories/reminiscence
  6. Exercising to music
  7. Breathing exercises and relaxing exercises
  The treatment is following the principles of resource oriented music therapy as described by Rolvsjord et al (2005)

SUMMARY:
This study evaluates the effect and process of individualized music therapy for home-dwelling persons with mild to moderate dementia. The music therapy is administered individually and includes a close caregiver. Memory of familiar music is found to be retained in persons with dementia. It is assumed to facilitate autobiographical memories and stimulate interaction with significant others. Based on time series analyses we will use statistical process control to evaluate when and how change occur.

DETAILED DESCRIPTION:
Dementia is often followed by complicating symptoms such as anxiety, depression, agitation, hallucination and sleep disorders. The progression of dementia can threaten the relationship between the person with dementia (PWD) and their relatives. One reason is the possible loss of reciprocity and a mutual supportive relationship. This may influence the quality of life in both the PWD and their relatives and increase the caregiver-burden. The music therapy in this intervention is focusing on increasing positive emotions, increasing reciprocity and stimulating communication.

The 1st, 5th and 10th music therapy-session is video-recorded. The first 5 recorded minutes before the sessions will provide a baseline of the observed primary outcomes throughout the session. Videos are analyzed to examine changes in social communication behavior and emotional well-being. Time-series analysis of the observations will be conducted, enabling us to evaluate potential effects of the therapeutic interventions and to find out when, why and to what extent changes unfold in real time. The pre-post measures are secondary. The project is a merging and further development of two recent music therapy designs. (Articles cited in the references.)

ELIGIBILITY:
Inclusion Criteria:

* The patient is diagnosed with Dementia of the Alzheimer's type, Vascular Dementia, Dementia with Lewy bodies, Parkinsons's Disease Dementia (ICD-10 criteria)
* The severity of the cognitive impairment is within the range of 0,5 - 2 when assessed with The Clinical Dementia Rating Scale (CDR)
* A caregiver chosen by the patient commits to involvement in the treatment as a collateral (i.e. spouse, child, grandchild, sibling, close friend)
* Use of psychotropic medication has been stable during the past 2 weeks
* The PWD is able to answer simple self-report questionnaires on their own or when interviewed by a trained professional
* Informed consent is obtained from patients and caregiver
* The PWD's are living in their home, in assisted living facilities or only periodical living in care homes.

Exclusion Criteria:

* Severe dementia(a score of 3> on CDR).
* Severe aphasia
* Frontotemporal dementia
* Comorbid diagnosis of bipolar disorder, diagnosis of schizophrenia and related disorders
* Changes in psychotropic medications in the past 2 weeks. If so, the medication needs to be stable before pre-assessment is undertaken
* Severe psychotic symptoms or serious risk of suicide
* Permanent living arrangement in nursing home, or planned temporary stay during the treatment period

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in social interaction behavior throughout the music therapy session compared to baseline(Verbal and Nonverbal Interaction Scale (VNVIS)) | Baseline (the first 5 videorecorded minutes before the music therapy) up to 45 minutes with music therapy intervention. The 1st, 5th and 10th session is videorecorded. Observation-interval is 30 seconds.
  Verbal and nonverbal interaction scale(VNVIS) is a standardized observational instrument for assessing prosocial and nonsocial verbal and nonverbal communication behavior between a person with dementia and their close caregiver. The scale is measuring both prosocial and nonsocial behavior, 26 items, 13 pr subscale. The person can score from 0-13 points on prosocial items pr timepoint, higher score indicates more prosocial behavior is present. The same holds for nonsocial behavior, the higher score indicates more nonsocial behavior observed.
Observable signs of well being (OSWDS) | Baseline (the first 5 videorecorded minutes before the music therapy) up to 45 minutes with music therapy intervention. The 1st, 5th and 10th session is videorecorded. Observation-interval is 30 seconds.
  The observable signs of wellbeing in dementia- scale (OSWDS) is a scale for proxy-rated well being in persons with dementia. The scale is under development, and is tested during the intervention. It consists of 10 items measuring from 0-10 points. Each item is rated as present or non-present during the time interval. Higher score indicates higher levels of observed wellbeing.
Change in self reported mood before and after the music therapy session (Visual Analogue Mood Scale (VAMS)) | Assessment before and after every music therapy session (10 weeks) and before and after every musical activity with the relative (10 weeks)
  VAMS is a standardized visual analogue scale tailored to persons with cognitive impairment measuring 8 self reported mood states. Each state is scored by marking on a 10 cm line by the person with dementia. The score is calculated by measuring the point on the line in mm, and the range is 0-100, were 100 indicates maximum emotional experience.

SECONDARY OUTCOMES:
Change in Neuropsychiatric symptoms (NPI-Q) | Baseline and post-treatment (up to two weeks after the intervention period)
  NPI-Q is a standardized measure of common neuropsychiatric symptoms following dementia. The scale consists of 12 items rated from 0-3. Items are summed, and the range is 0-36. Higher score means more severe neuropsychiatric symptoms.
Change in Quality of life in Alzheimer Dementia (QoL-AD) | Baseline and post-treatment (up to two weeks after the intervention period)
  QoL-AD is a standardized interview designed to measure items concerning the experienced quality of life in persons with dementia. The scale consists of 15 items from 1-4. The items are summed, and the range is 15-60. Higher score means higher self-reported quality of life.
Change in Relative Stress Scale (RSS) | Baseline and post-treatment (up to two weeks after the intervention period)
  RSS is a standardized measure of self-reported caregiver burden in carers of PWD. 15 items are scored from 0-4, giving a range from 0-60. A higher score indicates more severe stress for the caregiver.
Change in Music in Dementia Assessment Scales (MiDAS) | Before and after every music therapy session (10 weeks)
  MiDAS is a standardized music therapy outcome scale measuring clinical response to the intervention. The scale consists of 5 items on a visual analogue scale, and the music therapist score the items for the 5 first minutes and for the 5 most significant minutes in the session. Each item has a range from 0-100, were a higher score means a higher level of involvement in the music therapy. The 5 items are reviewed separately.

OTHER OUTCOMES:
Mini Mental Status Examination (MMSE) | Baseline
  Screening instrument for cognitive impairment. The scale consists of 30 questions and tasks. The range is 0-30 points, were a higher score indicates higher cognitive functions.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Hilde Nordhus, Professor, PhD, Principal Investigator — University of Bergen
Locations (1):
- NKS Olaviken Alderspsykiatriske sykehus, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shall A, Haberstroh J, Pantel J. Time series analysis of individual music therapy in dementia. Effects on communication behavior and emotional well-being. Gero Psych 28 (3): 113-122, 2015
- [Background] Baker FA, Grocke D, Pachana NA, Clair AA. Connecting through music: a study of a spousal caregiver-directed music intervention designed to prolong fulfilling relationships in couples where one person has dementia. Australian Journal of Music Therapy, 23: 4-21, 2012.
- [Background] Rolvsjord R, Gold C, Stige B. Research rigour and therapeutic flexibility: Rationale for a therapy manual developed for a randomised controlled trial. Nordic Journal of Music Therapy 14(1), 15-32, 2005.